CLINICAL TRIAL: NCT00098839
Title: A Feasibility Pilot and Phase II Study Of Chemoimmunotherapy With Epratuzumab (IND #12034) for Children With Relapsed CD22-Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Chemoimmunotherapy With Epratuzumab in Relapsed Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL04P2; NCI-2011-01624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL04P2 (Other: Children's Oncology Group); CDR0000396777 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Recurrent Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; palmitoyl-L-asparaginase; Doxorubicin; Hydrocortisone; Vincristine; epratuzumab; Cytarabine; Prednisone; pegaspargase; Dexrazoxane; Razoxane; Methotrexate; merphos; Etoposide; Cyclophosphamide; Leucovorin; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reinduction Chemoimmunotherapy with Epratuzumab once weekly (Experimental): Four weekly doses of epratuzumab (360 mg/m2/dose) IV days 1, 8, 15, 22. Also received vincristine sulfate, prednisone, pegaspargase, doxorubicin hydrochloride, dexrazoxane hydrochloride, etoposide, cyclophosphamide, filgrastim, high-dose (HD) methotrexate with Leucovorin calcium rescue, L-asparaginase, cytarabine, IT cytarabine, IT methotrexate (CNS-negative), Intrathecal triple therapy (ITT) (methotrexate, cytarabine, therapeutic hydrocortisone for CNS-positive) during the 3 blocks of reinduction therapy.
  Interventions: Drug: L-asparaginase; Drug: doxorubicin hydrochloride; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Biological: epratuzumab; Drug: cytarabine; Drug: prednisone; Drug: pegaspargase; Drug: dexrazoxane hydrochloride; Drug: methotrexate; Drug: etoposide; Drug: cyclophosphamide; Drug: leucovorin calcium; Biological: filgrastim
- Reinduction Chemoimmunotherapy with Epratuzumab twice weekly (Experimental): Eight 8 twice-weekly doses of epratuzumab (360 mg/m2/dose) IV days 1, 4, 8, 11, 15, 18, 22 & 25. Also received vincristine sulfate, prednisone, pegaspargase, doxorubicin hydrochloride, dexrazoxane hydrochloride, etoposide, cyclophosphamide, filgrastim, high-dose (HD) methotrexate with Leucovorin calcium rescue, L-asparaginase, cytarabine, IT cytarabine, IT methotrexate (CNS-negative), Intrathecal triple therapy (ITT) (methotrexate, cytarabine, therapeutic hydrocortisone for CNS-positive) during the 3 blocks of reinduction therapy.
  Interventions: Drug: L-asparaginase; Drug: doxorubicin hydrochloride; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Biological: epratuzumab; Drug: cytarabine; Drug: prednisone; Drug: pegaspargase; Drug: dexrazoxane hydrochloride; Drug: methotrexate; Drug: etoposide; Drug: cyclophosphamide; Drug: leucovorin calcium; Biological: filgrastim

INTERVENTIONS:
Drug: L-asparaginase — Given IM
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: therapeutic hydrocortisone — 40 mg/m2/day PO divided BID or TID
  Other Names: Aeroseb-HC; Barseb HC; Cetacort; Cort-Dome; Cortef
Drug: vincristine sulfate — Given IV
  Other Names: liposomal vincristine; Marqibo; vincristine liposomal; vincristine sulfate liposome injection
Biological: epratuzumab — Given IV
  Other Names: AMG 412; LL2; MOAB LL2; monoclonal antibody LL2
Drug: cytarabine — Given IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Drug: pegaspargase — Given IM
  Other Names: L-asparaginase with polyethylene glycol; Oncaspar; PEG-ASP; PEG-L-asparaginase
Drug: dexrazoxane hydrochloride — Given IV
  Other Names: Cardioxane; Savene; Totect; Zinecard
Drug: methotrexate — Given IT
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen

SUMMARY:
This Phase II trial is studying how well giving epratuzumab together with an established chemotherapy platform works in treating young patients with relapsed acute lymphoblastic leukemia. Monoclonal antibodies, such as epratuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing them or by stopping them from dividing. Giving monoclonal antibody therapy in combination chemotherapy may kill cancer cells more effectively.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of epratuzumab administered alone and in combination with re-induction combination chemotherapy in pediatric patients with relapsed CD22-positive acute lymphoblastic leukemia.

II. Determine the toxic effects of this regimen in these patients.

III. Determine the antitumor activity of this regimen in these patients.

IV. To estimate the remission re-induction rate and four-month event-free survival (EFS) for patients with early first relapse ALL who receive epratuzumab in combination with cytotoxic thermotherapy.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of epratuzumab in these patients. II. Determine the biologic activity of epratuzumab using measurements of minimal residual disease in these patients.

III. Determine the human anti-human antibody (HAHA) response in patients treated with this regimen.

OUTLINE: This is a multicenter study comprising a feasibility part A (closed to accrual as of 10/30/06) followed by a pilot part B study. A Simon's two stage design was initially used to evaluate the efficacy of the once weekly dosing schedule for part B patients (called B1 cohort), which planned to accrue a total of 112 patients with 56 to be enrolled at the first stage. After completion the accrual of stage 1, i.e. after 56 patients were enrolled, the design of part B was revised to evaluate a modified doing schedule (twice weekly doing, called B2 cohort) using a stratified two-stage design by London and Chang (2005), where patients enrolled to B2 were stratified according to relapse (first early marrow relapsed occurring < 18 months from initial diagnosis vs 18-36 months from initial diagnosis).

PART A (CLOSED TO ACCRUAL 10/30/06):

REDUCTION THERAPY: Patients receive epratuzumab IV over several hours on days -14, -10, -6, and -2 and cytarabine intrathecally (IT) on day -14*.

NOTE: *Patients who receive IT chemotherapy within 7 days of study entry as prior maintenance chemotherapy (e.g., before the diagnosis of relapse) did not receive this first dose of IT cytarabine.

RE-INDUCTION THERAPY (BLOCK 1): Patients received vincristine IV on days 1, 8, 15, and 22; oral prednisone two or three times daily on days 1-29; pegaspargase intramuscularly (IM) on days 2, 9, 16, and 23; dexrazoxane IV followed by doxorubicin IV over 15 minutes on day 1; methotrexate IT on days 15 and 29 for CNS-negative disease; and epratuzumab IV over 1 hour on days 8, 15, 22, and 29. Patients with CNS-positive disease also received triple IT therapy (ITT) consisting of methotrexate, cytarabine, hydrocortisone on days -10, -6, 1 and 15.

RE-INDUCTION THERAPY (BLOCK 2): Beginning at least 7 days after the last dose of IT chemotherapy, patients received etoposide IV over 2 hours and cyclophosphamide IV over 30 minutes on days 1-5. Patients also received high-dose methotrexate IV continuously over 24 hours on day 22. Beginning 42 hours after the start of the methotrexate infusion (day 24), patients received leucovorin calcium IV every 6 hours for a minimum of 3 doses. Patients with CNS-negative disease also receive methotrexate IT on days 1 and 22. Patients with CNS-positive disease will receive triple IT as in re-induction therapy (block 1) on days 1 and 22. Patients received filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 6 and continuing until blood counts recover.

RE-INDUCTION THERAPY (PART 3): Beginning at least 7 days after the last dose of IT chemotherapy, patients received cytarabine IV over 3 hours twice daily on days 1, 2, 8, and 9 and native E. Coli asparaginase IM on days 2 and 9. Patients receive G-CSF SC once daily beginning on day 10 and continuing until blood counts recovered.

PART B:

RE-INDUCTION THERAPY (BLOCK 1): Patients received vincristine, prednisone, pegaspargase, doxorubicin, cytarabine, methotrexate, and epratuzumab as in phase I re-induction therapy (block 1). Epratuzumab was given on Days 1, 8, 15 and 22 before amendment 5 (B1 cohort) and on Days 1, 4, 8, 11, 15, 18, 22 and 25 after amendment 5 (B2 cohort) Patients with CNS-negative disease received methotrexate IT on days 1 and 22. Patients with CNS-positive disease received triple IT therapy comprising methotrexate, cytarabine, and hydrocortisone on days 8, 15, 22, and 29.

RE-INDUCTION THERAPY (BLOCKS 2 AND 3): Patients received re-induction therapy blocks 2 and 3 as in the part A re-induction therapy (blocks 2 and 3) portion of the study.

Patients are followed annually.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B lymphoblastic leukemia (B-ALL)

  * At least 25% expression of CD22 by immunophenotyping
  * In marrow relapse (M3 bone marrow) with or without associated extramedullary disease as defined by 1 of the following:

    * In first or later marrow relapse occurring any time after initial diagnosis (part A [closed to accrual as of 10/30/06] or B)
    * In first, early marrow relapse with or without associated extramedullary disease occurring < 36 months from the time of initial diagnosis (part B only)
* No B-cell L3 morphology OR evidence of a regulator gene that codes for a transcription factor (MYC) translocation by molecular or cytogenetic analysis
* No Down syndrome
* Patients with CNS or other extramedullary site involvement are allowed
* Performance status - Karnofsky 50-100% (for patients > 10 years of age)
* Performance status - Lansky 50-100% (for patients ≤ 10 years of age)
* White Blood Count (WBC) ≤ 50,000/mm^3 (part A only [closed to accrual as of 10/30/06])
* Bilirubin ≤ 1.5 times upper limit of normal unless disease-related (ULN)
* Alanine aminotransferase (ALT) ≤ 5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine clearance OR radioisotope glomerular filtration rate ≥ 70 mL/min
* Creatinine as defined by age as follows:

  * ≤ 0.5 mg/dL (for patients < 1 year old)
  * ≤ 0.8 mg/dL (for patients 1 to 5 years old)
  * ≤ 1.0 mg/dL (for patients 6 to 10 years old)
  * ≤ 1.2 mg/dL (for patients 11 to 15 years old)
  * ≤ 1.5 mg/dL (for patients > 15 years old)
* Shortening fraction ≥ 27% by echocardiogram
* Ejection fraction ≥ 45% by Multi Gated Acquisition Scan (MUGA)
* No dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94%
* No active or uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Recovered from prior immunotherapy
* At least 4 months since prior stem cell transplantation or rescue AND no evidence of active graft-vs-host disease
* At least 7 days since prior hematopoietic growth factors
* At least 7 days since prior biologic therapy*
* No other concurrent immunotherapy
* No other concurrent biologic therapy
* Recovered from prior chemotherapy

  * No waiting period for children who relapse while receiving standard ALL maintenance therapy
* No prior cumulative anthracycline exposure > 400 mg/m^2*
* No concurrent chemotherapy
* Recovered from prior radiotherapy
* No concurrent radiotherapy
* At least 2 days since prior hydroxyurea
* No other concurrent investigational drugs
* No other concurrent anticancer agents

Ages: 2 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2005-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raetz, MD, Principal Investigator — Children's Oncology Group
Locations (46):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Hospital Sainte-Justine, Montreal, Quebec, Canada
- San Jorge Children's Hospital, Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The phase I part of the study was completed as of August 2006. The study was amended on 11/10/2006 and Part B (phase 2 pilot) was opened on 01/08/2007 which consisted of two dosing schedules for epratuzumab: weekly for four doses during Block 1 and twice weekly for eight doses during Block 1. This report is limited to Part B (116 enrollments).
Period: Overall Study
Arm/Group | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly
Started | 56 | 60
Completed | 24 | 27
Not Completed | 32 | 33
Not completed — Adverse Event | 5 | 2
Not completed — Death | 1 | 2
Not completed — Physician Decision | 4 | 14
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Refusal of further protocol therapy | 3 | 1
Not completed — Relapse | 6 | 3
Not completed — M2/M3 marrow on Day 15 of Block 2 | 10 | 11
Not completed — Ineligible | 2 | 0

BASELINE CHARACTERISTICS:
Population: Ineligible patients (2) are not included in baseline population.
Groups:
- Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly: Four weekly doses of epratuzumab (360 mg/m2/dose) IV days 1, 8, 15, 22. Also received vincristine sulfate, prednisone, pegaspargase, doxorubicin hydrochloride, dexrazoxane hydrochloride, etoposide, cyclophosphamide, filgrastim, HD methotrexate with Leucovorin calcium rescue, L-asparaginase, cytarabine, IT cytarabine, IT methotrexate (CNS-negative), ITT (methotrexate, cytarabine, therapeutic hydrocortisone for CNS-positive) during the 3 blocks of reinduction therapy.
  L-asparaginase: Given IM
  doxorubicin hydrochloride: Given IV
  therapeutic hydrocortisone: 40 mg/m2/day PO divided BID or TID
  vincristine sulfate: Given IV
  epratuzumab: Given IV
  cytarabine: Given IT
  prednisone: Given orally
  pegaspargase: Given IM
  dexrazoxane hydrochloride: Given IV
  methotrexate: Given IT
  etoposide: Given IV
  cyclophosphamide: Given IV
  leucovorin calcium: Given IV
  filgrastim: Given SC
- Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly: Eight 8 twice-weekly doses of epratuzumab (360 mg/m2/dose) IV days 1, 4, 8, 11, 15, 18, 22 & 25. Also received vincristine sulfate, prednisone, pegaspargase, doxorubicin hydrochloride, dexrazoxane hydrochloride, etoposide, cyclophosphamide, filgrastim, HD methotrexate with Leucovorin calcium rescue, L-asparaginase, cytarabine, IT cytarabine, IT methotrexate (CNS-negative), ITT (methotrexate, cytarabine, therapeutic hydrocortisone for CNS-positive) during the 3 blocks of reinduction therapy.
  L-asparaginase: Given IM
  doxorubicin hydrochloride: Given IV
  therapeutic hydrocortisone: 40 mg/m2/day PO divided BID or TID
  vincristine sulfate: Given IV
  epratuzumab: Given IV
  cytarabine: Given IT
  prednisone: Given orally
  pegaspargase: Given IM
  dexrazoxane hydrochloride: Given IV
  methotrexate: Given IT
  etoposide: Given IV
  cyclophosphamide: Given IV
  leucovorin calcium: Given IV
  filgrastim: Given SC
- Total: Total of all reporting groups
Arm/Group | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly | Total
Number analyzed (Participants) | 54 | 60 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (5.54) | 9.7 (5.44) | 10.1 (5.48)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 55 | 103
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 52
  Male | 31 | 31 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 6 | 16
  White | 38 | 46 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 20 | 34
  Not Hispanic or Latino | 37 | 38 | 75
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Remission Re-induction (CR2) Rate
Description: The proportion of patients who achieved complete response at the end Block 1 of re-induction therapy. Complete Remission (CR) - Attainment of M1 bone marrow (<5% blasts) with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral counts (ANC >1000/uL and platelet count >100,000/uL). Partial Remission (PR) - Complete disappearance of circulating blasts and achievement of M2 marrow status (5% or < 25% blast cells and adequate cellularity). Partial Remission Cytolytic (PRCL) - Complete disappearance of circulating blasts and achievement of at least 50% reduction from baseline in bone marrow blast count. Minimal Response Cytolytic (MRCL) - 50% reduction in the peripheral blast count with no increase in peripheral white blood cell count.
Time Frame: At the end of Block 1 of re-induction therapy (day 36)
Population: Evaluable patients at the end of Block 1. There were 2 ineligible patients for once weekly arm and 6 patients not evaluable at the end of block 1 re-induction therapy. There were 10 patients for twice weekly arm not evaluable at the end of block 1 re-induction therapy.
Measure: Number; unit: proportion of participants
Arm/Group | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly
Number analyzed (Participants) | 48 | 50
proportion of participants | .646 | .660

2. Primary Outcome: Event-free Survival Rate
Description: Proportion of patients who were event free at 4 months
Time Frame: At 4 months after enrollment
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly
Number analyzed (Participants) | 48 | 50
Proportion of participants | .604 | .640

3. Primary Outcome: Rate of Minimal Residual Disease (MRD) < 0.01%
Description: Proportion of patients (evaluable and had MRD measured at the end of Block 1) who had MRD < 0.01%.
Time Frame: At the end of Block 1 of re-induction therapy (day 36)
Population: Evaluable patients who had MRD measured at the end of Block 1. There were 2 ineligible patients for once weekly arm and 13 patients where MRD was not measured at the end of block 1 re-induction therapy. There were 16 patients for twice weekly arm where MRD was not measured at the end of block 1 re-induction therapy.
Measure: Number; unit: Proportion of participants
Arm/Group | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly
Number analyzed (Participants) | 41 | 44
Proportion of participants | .195 | .295

4. Secondary Outcome: Pharmacokinetics
Description: Mean trough serum concentration measured before final dose of epratuzumab.
Time Frame: Up to day 36
Population: Pharmacokinetics (PK) were added to the protocol with amendment 5A for the twice weekly dosing schedule of Epratuzumab. Hence, PK studies were limited to evaluable patients on this Arm only.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Twice Weekly Dosing Schedule: Epratuzumab 360 mg/m2 x 8 doses - Part B (Amendment 5)
Arm/Group | Twice Weekly Dosing Schedule
Number analyzed (Participants) | 26
ug/mL | 501 (149)

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Ineligible patients (2) are not included in adverse event reporting for the once weekly arm.
Arm/Group | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly
Serious Adverse Events (participants affected / at risk) | 16/54 | 20/60
Other Adverse Events (participants affected / at risk) | 44/54 | 41/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly (N=54) | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly (N=60)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 11 (11)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 16 (21) | 20 (21)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 4 (4) | 0 (0)
GGT increased (Investigations) | 3 (3) | 0 (0)
INR increased (Investigations) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 5 (5) | 4 (4)
Lymphocyte count decreased (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 2 (2)
Platelet count decreased (Investigations) | 4 (5) | 2 (2)
Serum amylase increased (Investigations) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 5 (5) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 4 (4) | 3 (3)
Vascular disorders - Other (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reinduction Chemoimmunotherapy With Epratuzumab Once Weekly (N=54) | Reinduction Chemoimmunotherapy With Epratuzumab Twice Weekly (N=60)
Anemia (Blood and lymphatic system disorders) | 36 (45) | 41 (49)
Febrile neutropenia (Blood and lymphatic system disorders) | 18 (18) | 22 (23)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Eye disorders - Other (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (2)
Irritability (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 4 (4)
Anaphylaxis (Immune system disorders) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 3 (3) | 3 (3)
Infections and infestations - Other (Infections and infestations) | 28 (29) | 19 (20)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 8 (8) | 15 (16)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 9 (9) | 11 (12)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Fibrinogen decreased (Investigations) | 2 (2) | 5 (5)
GGT increased (Investigations) | 3 (3) | 1 (1)
Lipase increased (Investigations) | 6 (6) | 4 (4)
Lymphocyte count decreased (Investigations) | 10 (15) | 22 (29)
Neutrophil count decreased (Investigations) | 38 (43) | 40 (42)
Platelet count decreased (Investigations) | 39 (54) | 38 (46)
Serum amylase increased (Investigations) | 3 (3) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 34 (44) | 40 (44)
Acidosis (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (20) | 15 (15)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (10) | 8 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 16 (16) | 16 (19)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 11 (11) | 9 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Arachnoiditis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 2 (2)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.